CLINICAL TRIAL: NCT02586597
Title: Paired Associative Stimulation Modulates Motor Excitability and Plasticity in Chronic Stroke Patients
Brief Title: Paired Associative Stimulation in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Xingbao Li, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Device Feasibility
Other Study IDs: Pro00040369
Record Dates: First submitted 2015-03-17; First posted 2015-10-26 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-02

CONDITIONS: Stroke
Keywords: Stroke; PAS; TMS; cortical excitability; plasticity
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PAS 10: TMS and median nerve stimulation (Experimental): Paired associative stimulation (PAS) is a new technique where one pairs a peripheral stimulation with centrally applied transcranial magnetic stimulation (TMS), and produces plasticity, as measured by TMS MEP's. Currently PAS is performed with median nerve stimulation. The interval between median nerve stimulation and TMS was chosen to be 10 ms, which is called PAS10. PAS 10: TMS and median nerve stimulation: 240 paired median nerve stimulation and TMS during 20 minutes.
  Interventions: Device: Transcranial magnetic stimulation & median nerve stimulation
- PAS 25:TMS and median nerve stimulation (Experimental): PAS 25: The interval between median nerve stimulation and TMS was chosen to be 25 ms, which is called PAS25. PAS 25:TMS and median nerve stimulation: 240 paired median nerve stimulation and TMS during 20 minutes.
  Interventions: Device: Transcranial magnetic stimulation & median nerve stimulation
- PAS100:TMS and median nerve stimulation (Sham Comparator): PAS Control Paradigm: The interval between median nerve stimulation and TMS was chosen to be 100 ms, which is called PAS100. PAS100:TMS and median nerve stimulation: 240 paired median nerve stimulation and TMS during 20 minutes.
  Interventions: Device: Transcranial magnetic stimulation & median nerve stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation & median nerve stimulation — Paired associative stimulation (PAS) is a new technique where one pairs a peripheral stimulation with centrally applied transcranial magnetic stimulation (TMS), and produces plasticity, as measured by TMS MEP's. Currently PAS is performed with median nerve stimulation.
  PA25: The interval between median nerve stimulation and TMS was chosen to be 25 ms, which is called PAS25. 240 paired TMS and median nerve stimulation at a frequency of 0.2 Hz over 20 min.
  PAS10: 240 paired TMS and median nerve stimulation with interval of 10 min second at a frequency of 0.2 Hz over 20 min.
  PAS100: 240 paired TMS and median nerve stimulation with interval of 100 min second at a frequency of 0.2 Hz over 20 min.

SUMMARY:
Stroke is the third most common cause of death in the United States after heart disease and cancer, and the leading cause of long-term disability. This work will develop an innovative brain stimulation method (paired associative stimulation) which might set the stage for a new treatment for stroke rehabilitation.

DETAILED DESCRIPTION:
Stroke is the third most common cause of death in the United States after heart disease and cancer. An innovative recovery treatment is in demand for stroke motor recovery. Paired associative stimulation (PAS) is a new technique where one pairs a peripheral stimulation with centrally applied transcranial magnetic stimulation (TMS), and produces plasticity, as measured by TMS motor-evoked potentials (MEP's). The investigators will also compare post-stroke patients to healthy controls on the modulation effect of PAS and motor behavior measures.

Aim1. To investigate whether PAS (PAS25 or PAS10) can modulate motor excitability and plasticity;

Aim2. To investigate whether PAS can modify motor behaviors measures in both post-stroke patients and healthy controls;

Aim3. To investigate whether post-stroke patients show different modulation of PAS on both cortical plasticity and motor behavior measure compared to healthy controls.

For this study the investigators will enroll a total of 10 chronic stroke patients and 10 neurologically healthy controls matched for age and gender. Participants will have 4 visits. The first visit is for screening. They will receive either sham PAS or real PAS25 or real PAS10 at each following treatment visit.

Experimental Methods: Clinical Behavioral Measures: Handgrip; Nine-hole Peg Test; Wolf Motor Function Test; Imaging protocol: T1 weighted anatomical image, fluid attenuation inversion recovery (FLAIR) and diffusion tensor imaging (DTI); Stimulation locations: Left primary motor (M1); right median nerve; PAS methods: TMS stimulation will be delivered at 25 ms or 10 ms or 100 ms after median nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. first-ever ischemic stroke involving only one hemisphere;
3. Patient demonstrates at least 10 degrees of voluntary finger, thumb and wrist extension; ;
4. 6 - 24 months after ischemic stroke

Exclusion Criteria:

1. Primary or secondary intracerebral hematoma, or subarachnoid hemorrhage, or subdural/epidural hematoma;
2. Bihemispheric ischemic strokes;
3. History of prior stroke or old infarct demonstrated on the CT or MRI or documented in medical records or current on anticoagulant;
4. Other concomitant neurological disorders, such as brain tumor, abscess or spinal cord disease affecting upper extremity motor function;
5. Documented history of dementia prior to index event;
6. Presence of any MRI/TMS risk factors such as (a) an electrically, magnetically or mechanically activated implant including cardiac pacemaker, intracerebral vascular clips or any other electrically sensitive support system; (b) non-fixed metal in any part of the body, including a previous metallic injury to eye [all jewelry will be removed during stimulation]; (c) pregnancy, since the effect of TMS on the fetus is unknown, females of child bearing age will have to undergo a pregnancy test to confirm eligibility; (d) history of seizure disorder or post-stroke seizures. This last exclusion criterion applies only to the modulation portion of the proposal; (e) median nerve is damaged

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Intracortical facilitation | 10-day treatment
  the peak magnitude of MEP

SECONDARY OUTCOMES:
Clinical behavioral measures-Handgrip | 10-day treatment
  hand grip strength
Nine-hole peg test | 10-day treatment
  screening tool to administer Portable assess finger dexterity and median nerve function
wolf motor function test | 10-day treatment
  To measure upper extremity motor ability through timed and functional tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Li X, Ricci R, Large CH, Anderson B, Nahas Z, George MS. Lamotrigine and valproic acid have different effects on motorcortical neuronal excitability. J Neural Transm (Vienna). 2009 Apr;116(4):423-9. doi: 10.1007/s00702-009-0195-z. Epub 2009 Feb 24. PMID 19238517